CLINICAL TRIAL: NCT04158804
Title: PROcalcitonin Impact on Antibiotic Reduction, adverSe Events and AVoidable healthcarE Costs
Brief Title: PROcalcitonin Impact on Antibiotic Reduction, adverSe Events and AVoidable healthcarE Costs (ProSAVE): A RCT
Acronym: ProSAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: BRAHMS GmbH (Unknown); Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Principal Investigator, Michael K. Mansour, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2019P000362
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pneumonia, Bacterial
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Procalcitonin algorithm+stewardship team (Experimental): antibiotic prescription guided by PCT values
  Interventions: Diagnostic Test: procalcitonin
- standard group (No Intervention): standard of care guided by current guidelines

INTERVENTIONS:
Diagnostic Test: procalcitonin — accuracy of procalcitonin as a diagnostic marker in guiding antibiotic therapy in patients with a lower respiratory tract infection
  Arms: Procalcitonin algorithm+stewardship team

SUMMARY:
Trials comparing PCT-guided antibiotic algorithms to standard management show a significant reduction in antibiotic exposure without an increase in mortality or treatment failure. Despite this strong evidence from multiple studies a recent prospective multicentric interventional trial in the US fell short of demonstrating antibiotic reductions by PCT-guided antibiotic management. Amongst other limitations the authors of that study concluded that successful implementation of PCT may require closer educational oversight. As such, this study will compare effectiveness and safety of antibiotic prescription guided by a PCT-algorithm via a Stewardship Team over standard guidelines in hospitalized adult patients with suspected or confirmed LRTI (including sepsis with respiratory focus).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult patients ≥ 18 years of age
* Suspected or confirmed pneumonia <28 days at time of admission to the hospital (ED) who are prescribed antibiotics
* Minimum of 2 (two) blood samples available for PCT value assessment within 24 hours of hospitalization

Exclusion Criteria:

* Patient has tested positive for SARS-CoV-2
* Non-hospitalized patients
* Patients admitted to home health
* Major surgeries, defined as any procedure in which an incision is made with the exception of superficial procedures (eyes, cornea, skin, dental procedures), organs removed, or normal anatomy altered (e.g. open thoracic, abdominal and/or major orthopedic surgery), in the past 1 month or expected surgical procedure or patient receiving antibiotics for surgical prophylaxis
* Active metastatic cancer or neuroendocrine tumor or liquid tumor and/or on check point inhibitors within 3 months or has signs of mucositis (e.g. mouth lesions or intestinal bleeding)
* Known pregnancy
* Primary and acquired cell-mediated immune deficiency (HIV with CD4 <350 cells/mm³; receipt of systemic chemotherapy and/or biologics in the past 3 months for reasons other than malignancy)
* Infection where long course antibiotics are the standard of care(>2 weeks) other than anti-inflammatory reasons.
* Neutropenia (<1,500 ANC)
* Concomitant non-pulmonary bacterial infection that requires antibiotic therapy based on an active medical team decision
* Antibiotics given for non-infectious indications (e.g. rifaximin for hepatic encephalopathy)
* Patients with cystic fibrosis
* Patients receiving dialysis
* Patients with solid organ transplant, bone marrow transplant or stem cell transplant recipient
* ST elevation myocardial infarction
* Prior enrollment into this study within 30 days
* Patient experiencing major trauma defined as any injury that could cause prolonged disability and/or an Injury Severity Score >15, and/or burns or patient under extracorporeal circulation confirmed by a second research staff member.
* Patient with acute viral hepatitis and/or decompensated severe liver cirrhosis (Child-Pugh Class C).
* Patient with prolonged or severe cardiogenic shock, defined as decreased cardiac output leading to end organ injury (e.g. severe hypotension or AKI or oliguria or altered mental status or cool extremities or respiratory distress AND evidence of metabolic acidosis on lab testing)
* Patient with pancreatitis, chemical pneumonitis or heat stroke
* Active infection with invasive fungal pathogen (e.g. candidiasis, aspergillosis) or plasmodium falciparum malaria or mycobacteria
* Patient under treatment with OKT3 antibodies, OK-432, interleukins, TNF-alpha and other drugs stimulating the release of pro-inflammatory cytokines or resulting in anaphylaxis.
* Patient is under hospice care
* Patient with ventilator associated pneumonia
* Patients with untreated, active, and symptomatic autoimmune disease
* Patients with empyema, abscess, or cavitary/necrotizing pneumonia
* Patients actively enrolled in other clinical trial involving immunomodulatory therapy

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Mansour, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Charlotte Hungerford Hospital, Torrington, Connecticut
  - Grady Memorial Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Martha's Vineyard Hospital, Oak Bluffs, Massachusetts
  - North Shore Medical Center, Salem, Massachusetts
  - Texas Health Harris Methodist Hospital, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SOC): PCT results were hidden from the medical record and no ASP recommendation given.
- PCT/ASP: PCT results were posted in the medical record and ASP emailed recommendation to the medical team.
Period: Overall Study
Arm/Group | Standard of Care (SOC) | PCT/ASP
Started | 357 | 343
Completed | 357 | 343
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | PCT/ASP | Total
Number analyzed (Participants) | 357 | 343 | 700
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [61 to 84] | 71 [60 to 81] | 72 [61 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 164 | 330
  Male | 191 | 179 | 370
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 29 | 72
  Not Hispanic or Latino | 305 | 303 | 608
  Unknown or Not Reported | 9 | 11 | 20
Pneumonia Type [Count of Participants; unit: Participants]
  CAP (community-acquired pneumonia) | 205 | 196 | 401
  HCAP (healthcare-associated pneumonia) | 10 | 15 | 25
  Aspiration | 89 | 82 | 171
  Other | 53 | 50 | 103
Pneumonia Severity Index (PSI) [Count of Participants; unit: Participants] — The Pneumonia Severity Index is a clinical tool used to assess the severity of pneumonia based on several clinical factors, including demographics, comorbidities, physical exam findings, vital signs, and lab and imaging results.
  Participants
    Class I (lowest severity) | 14 | 16 | 30
    Class II | 45 | 44 | 89
    Class III | 78 | 64 | 142
    Class IV | 144 | 156 | 300
    Class V (highest severity) | 76 | 63 | 139

OUTCOME MEASURES:

1. Primary Outcome: Short Treatment of Pneumonia
Description: Proportion of patients with short treatment of pneumonia with antibiotics (less than 4 days, "shortABx")
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) | PCT/ASP
Number analyzed (Participants) | 357 | 343
Participants | 47 | 87

2. Secondary Outcome: Composite Safety Adverse Event Rate
Description: Composite endpoints include: all-cause in-hospital mortality, all-cause mortality after discharge (as available), hospital readmission, septic shock (vasopressor use for > 1 hour), mechanical ventilation (via endotracheal tube), required dialysis, lung abscess/empyema/cavitation/necrotizing pneumonia
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) | PCT/ASP
Number analyzed (Participants) | 357 | 343
Participants | 72 | 90

3. Secondary Outcome: Antibiotic Exposure at Discharge
Description: Duration of antibiotics prescribed at discharge
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care (SOC) | PCT/ASP
Number analyzed (Participants) | 357 | 343
days | 0 [0 to 4] | 0 [0 to 2]

4. Secondary Outcome: Days of Therapy Per 1000 Patient Days
Description: Days of therapy per 1000 patient days (inclusive of antibiotics prescribed at discharge)
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: Days of Therapy Per 1000 Patient Days
Arm/Group | Standard of Care (SOC) | PCT/ASP
Number analyzed (Participants) | 357 | 343
Days of Therapy Per 1000 Patient Days | 1.25 [0.78 to 2.67] | 1.14 [0.67 to 2]

5. Secondary Outcome: Length of Stay
Description: Length of stay in hospital
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care (SOC) | PCT/ASP
Number analyzed (Participants) | 357 | 343
days | 4 [2 to 7] | 4 [3 to 7]

6. Secondary Outcome: ICU Admissions
Description: Number of Participants Admitted to the ICU
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) | PCT/ASP
Number analyzed (Participants) | 357 | 343
Participants | 43 | 49

7. Other Pre Specified Outcome: Clostridium Difficile Infection (CDI)
Description: Treatment or readmission for CDI until day 30 after enrollment
Time Frame: 30 days
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Healthcare Economic Endpoints
Description: Costs associated with primary hospitalization, readmission for CDI, and loss of function
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected starting at enrollment day until 30 days after enrollment.
Arm/Group | Standard of Care (SOC) | PCT/ASP
All-Cause Mortality (participants affected / at risk) | 19/357 | 17/343
Serious Adverse Events (participants affected / at risk) | 76/357 | 81/343
Other Adverse Events (participants affected / at risk) | 0/357 | 0/343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=357) | PCT/ASP (N=343)
Death (General disorders) | 19 (19) | 17 (17)
Septic Shock (Infections and infestations) | 11 (11) | 13 (13)
Mechanical Ventilation (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 13 (13)
Dialysis (Renal and urinary disorders) | 3 (3) | 0 (0)
Empyema (Infections and infestations) | 3 (3) | 6 (6)
Readmission (General disorders) | 47 (47) | 57 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT04158804/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT04158804/SAP_001.pdf